CLINICAL TRIAL: NCT03609151
Title: Effects of Stereotactic Body Radiotherapy and Surgery for Early-stage Hepatocellular Carcinoma: a Prospective,Randomized Controlled Trial
Brief Title: Stereotactic Body Radiotherapy and Surgery for Early-stage Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR2018001024
Record Dates: First submitted 2018-07-02; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hepatocellular Carcinoma; Hepatectomy; Stereotactic Body Radiotherapy
Keywords: Hepatocellular carcinoma; Early-stage liver cancer; Hepatectomy; Stereotactic body radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Surgical Procedures, Operative; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): laparoscopic hepatectomy (surgery)
  Interventions: Procedure: laparoscopic hepatectomy (surgery)
- group B (Experimental): stereotactic body radiotherapy (SBRT)
  Interventions: Radiation: stereotactic body radiotherapy

INTERVENTIONS:
Procedure: laparoscopic hepatectomy (surgery) — Patients receive laparoscopic hepatectomy.
  Arms: group A
Radiation: stereotactic body radiotherapy — Patients receive stereotactic body radiotherapy(SBRT)
  Arms: group B

SUMMARY:
The prognosis of small liver cancer (≤5 cm) with stereotactic body radiotherapy (SBRT) is encouraging, the 1-year local control rate has been reported to be 95-100%, 3-year local control rate about 91%, and 3-year overall survival rate around 70%. So far, there is no randomized controlled study comparing SBRT and surgical treatment for early-stage liver cancer. It is hoped that this study will further compare the efficacy of SBRT and surgery for early stage liver cancer.

DETAILED DESCRIPTION:
Early stage liver cancer, according to Milan criteria, are chose for this study. The patients are divided into two groups randomly. Patients in group A receive laparoscopic hepatectomy, group B patients receive SBRT.The 3-year progression free survival, 3-year local recurrence free survival, 3- year overall survival and other endpoints events were recorded and analyzed, to assess whether SBRT is non-inferior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above.
2. Clinical or pathological diagnosis of hepatocellular carcinoma, initial treatment (without surgery, radiotherapy, chemotherapy or targeted therapy).
3. Early-stage hepatocellular carcinoma meeting the Milan criteria: single lesion ≤ 5cm, or tumor number ≤ 3, maximum diameter ≤ 3cm, no major vascular invasion of portal vein, hepatic vein, inferior vena cava, no bile duct invasion, no lymph node and extrahepatic metastasis.
4. No serious blood system, heart, lung, liver, kidney dysfunction and immune deficiency.
5. The neutrophil count is at least 1.0*10^9/ml, and the platelet count is at least 50*10^9/ml. Hemoglobin is at least 80g/L.
6. Men or women with fertility are willing to take contraceptive measures during the trial.
7. Eastern Cooperative Oncology Group score 0-1 points.
8. Expected survival period > 3 months.
9. Voluntary participation and signing of informed consent.

Exclusion Criteria:

1. Patients who have undergone chemoradiation or targeted therapy for liver cancer.
2. Recent hematemesis due to portal hypertension.
3. Child-Pugh score ≥10 points.
4. Total bilirubin>70umol/L, aspartate aminotransferase (ALT), alanine aminotransferase (AST) exceed the upper limit of normal 3 times.
5. who was considered unsuitable for surgery after hepatobiliary and pancreas multidisciplinary treatment（MDT） meeting.
6. Patients undergoing major surgery within 1 month of study initiation
7. Patients with previous history of malignancy (excludes tumor-free survival after treatment of basal cell carcinoma of the skin and carcinoma of the cervix in situ for more than 3 years)
8. Researchers consider it inappropriate to participate in the test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From the date of surgery or the first fraction of SBRT until the date of first progression (local or distant), assessed up to 3 years
  The duration (months) between the date of surgery or the first fraction of SBRT until the date of first progression

SECONDARY OUTCOMES:
Local recurrence free survival | From the date of surgery or the first fraction of SBRT until the date of local recurrence, assessed up to 3 years
  The duration (months) between the date of surgery or the first fraction of SBRT until the date of local recurrence
Overall survival | From the date of surgery or the first fraction of SBRT until the date of death, assessed up to 3 years
  The duration (months) between the date of surgery or the first fraction of SBRT until the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China